CLINICAL TRIAL: NCT03842605
Title: Efficacy of Strength Training in Improving Elbow Range of Motion and Function in Adults With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Oleson, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09062
Record Dates: First submitted 2013-04-20; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hemophilia; Elbow Joint Contracture
MeSH Terms: conditions — Hemophilia A | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Strength training (Experimental)
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Strength training

SUMMARY:
This is a research study of adults with hemophilia that have limitations in elbow joint motion that is the result of bleeding into the joint.

People with hemophilia who have bleeding into their elbow joint may have limitations in elbow joint movement and pain in the joint. This research is being done to determine the effect a strength training program has on the amount of movement people with hemophilia and elbow joint disease have.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Oregon health and Science University Hemophilia treatment Center
* greater or equal to 18 years old
* Loss of elbow range of motion that is greater than or equal to 5 degrees

Exclusion Criteria:

* Present inhibitor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2019-02 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Elbow range of motion | measurements to be taken at 4 and 8 weeks after entering study
  measurement of change of range of motion over time frame

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States